CLINICAL TRIAL: NCT05945940
Title: Prognostic Significance of Preoperative Nutritional Status for Postoperative Acute Kidney Injury in Elderly Patients Undergoing Major Abdominal Surgery
Brief Title: Preoperative Nutritional Status and Postoperative Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Rao Sun (Other)
Responsible Party: Sponsor-Investigator, Rao Sun, Associate chief physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJH-20230608A
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
There is a high prevalence of postoperative acute kidney injury (AKI) in patients who undergo intra-abdominal surgery, and it is particularly common in the elderly. Identifying high-risk patients for postoperative AKI early can facilitate the development of preventive and therapeutic management strategies.

The goal of this retrospective study is to investigate the predictive value of preoperative nutritional status, as measured by three scoring systems - the geriatric nutritional risk index (GNRI), prognostic nutritional index (PNI), and controlling nutritional status (CONUT) score - on postoperative AKI in elderly patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 65 years
2. intra-abdominal procedures including gastric, colorectal, pancreatic, prostate, and urinary bladder surgeries, as well as abdominal exploration.
3. surgery duration lasting longer than 2 hours.

Exclusion Criteria:

1. patients with an American Society of Anesthesiologists (ASA) physical status V.
2. those with concurrent cardiac or renal surgeries.
3. those with end-stage renal disease (i.e. a glomerular filtration rate of 15 mL/min/1.73 m2 or receiving haemodialysis).
4. those did not have sufficient data required for nutritional evaluation or AKI evaluation.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) who underwent a major abdominal surgery under general anesthesia at Tongji Hospital between July 2018 and December 2021 were included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 2977 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Within 7 days after surgery
  In accordance with the KDIGO creatinine criteria: a serum creatinine increases of 26.5 mmol/L within 48 hours or 1.5 times baseline within 7 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rao Sun, Dr., Principal Investigator — Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China.
Locations (1):
- Rao Sun, Wuhan, China

IPD SHARING:
Plan to Share IPD: No